CLINICAL TRIAL: NCT02880878
Title: ENRICH: A Multi-center, Randomized, Clinical Trial Comparing Standard Medical Management to Early Surgical Hematoma Evacuation Using Minimally Invasive Parafascicular Surgery (MIPS) in the Treatment of Intracerebral Hemorrhage (ICH).
Brief Title: ENRICH: Early MiNimally-invasive Removal of IntraCerebral Hemorrhage (ICH)
Acronym: ENRICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nico Corporation (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DC-6010
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Intracerebral Hemorrhage; Cerebral Hemorrhage; Intracerebral Haemorrhage
Keywords: Subcortical Intracerebral Hemorrhage; Intracerebral Hemorrhage; Intracranial Hemorrhages; ICH; Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Pathologic Processes; MIPS; Minimally Invasive Parafascicular Surgery; Neurosurgery; Medical Economic; Hospital Economics
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Pathologic Processes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Surgical Hematoma Evacuation (Experimental): Subjects will receive early surgical hematoma evacuation using Minimally Invasive Parafascicular Surgery (MIPS).
  Interventions: Procedure: Early Surgical Hematoma Evacuation
- Medical Management (No Intervention): Subjects will receive standard of care medical management for ICH.

INTERVENTIONS:
Procedure: Early Surgical Hematoma Evacuation — Early Minimally Invasive Parafascicular Surgery (MIPS)
  Arms: Early Surgical Hematoma Evacuation

SUMMARY:
This is a multicenter, randomized, adaptive clinical trial comparing standard medical management to early (<24 hours) surgical hematoma evacuation using minimally invasive parafascicular surgery (MIPS) in the treatment of acute spontaneous supratentorial intracerebral hemorrhage.

DETAILED DESCRIPTION:
The ENRICH trial will compare the outcomes between early surgical intervention using the BrainPath® Approach (i.e., MIPS) and a medically managed cohort. The integrated surgical approach includes a combination of available technologies, including the FDA-cleared NICO BrainPath® for non-disruptive access and NICO Myriad® to achieve the goal of maximum clot evacuation. The medically managed cohort will be treated according the Clinical Standardization Guidelines (CSG) as adapted by Emory University from the 2015 AHA/ASA Guidelines for the Management of Spontaneous Intracerebral Hemorrhage. Clinical efficacy will be determined by demonstrating an improvement in functional outcome, as determined by a blinded-assessment of the 180-day utility-weighted modified Rankin Scale (mRS).

Data suggests improved mortality rates and potential functional benefits of surgical ICH evacuation. The methodology proposed for this trial was tested in a preliminary series of 39 patients treated for supratentorial spontaneous ICH and retrospectively reviewed (Labib et al.). These results were replicated in a single center retrospective series of 18 patients (Bauer et al.). Despite positive results of both studies and the widely accepted benefit of the BrainPath Approach (i.e., MIPS) for subcortical lesions, stronger evidence supporting the use of these techniques in ICH is needed for the technique to become universally validated.

CONTACTS:

Sponsor - Primary: Penny Sekerak, MBA, BA, RN (317) 569-1229, Penny.Sekerak@niconeuro.com

Sponsor - Backup: Jennifer Carroll, (317) 709-2466, Jennifer.Carroll@niconeuro.com

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Pre-randomization head CT demonstrating an acute, spontaneous, primary ICH
* ICH volume between 30 - 80 mL
* Study intervention can reasonably be initiated within 24 hours after the onset of stroke symptoms. If the actual time of onset is unclear, then the onset will be considered the time that the subject was last known to be well
* Glasgow Coma Score (GCS) 5 - 14
* Historical Modified Rankin Score 0 or 1

Exclusion Criteria:

* Ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, Moyamoya disease, venous sinus thrombosis, mass or tumor, hemorrhagic conversion of an ischemic infarct, recurrence of a recent (<1 year) ICH, as diagnosed with radiographic imaging
* NIHSS < 5
* Bilateral fixed dilated pupils
* Extensor motor posturing
* Intraventricular extension of the hemorrhage is visually estimated to involve >50% of either of the lateral ventricles
* Primary Thalamic ICH
* Infratentorial intraparenchymal hemorrhage including midbrain, pontine, or cerebellar
* Use of anticoagulants that cannot be rapidly reversed
* Evidence of active bleeding involving a retroperitoneal, gastrointestinal, genitourinary, or respiratory tract site
* Uncorrected coagulopathy or known clotting disorder
* Platelet count < 75,000, International Normalized Ratio (INR) > 1.4 after correction
* Patients requiring long-term anti-coagulation that needs to be initiated < 5 days from index ICH
* End stage renal disease
* Patients with a mechanical heart valve
* End-stage liver disease
* History of drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Positive urine or serum pregnancy test in female subjects without documented history of surgical sterilization or is post-menopausal
* Known life-expectancy of less than 6 months
* No reasonable expectation of recovery, Do-Not-Resuscitate (DNR), or comfort measures only prior to randomization
* Participation in a concurrent interventional medical investigation or clinical trial.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent
* Homelessness or inability to meet follow up requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Functional Improvement - mRS | 180 days
  Functional Improvement as determined by utility-weighted modified Rankin Scale (mRS) at 180-days

SECONDARY OUTCOMES:
Safety - Procedure-Related Mortality | 30 days
  Safety will be assessed by determining procedure-related mortality by comparing rates of mortality at 30 days for patients that underwent MIPS with medically treated patients
Safety - Hemorrhage Volume | 24 hours
  Safety will be assessed by evaluating whether MIPS does not result in an increase in hemorrhage volume between index CT and 24-hour follow-up CT as compared to medically treated patients
Economic | 30, 90, 120, and 180 days
  Economic differential as determined by quantification of the cost per quality-adjusted life-years (QALY) gained through MIPS

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Barrow, MD, Principal Investigator — 1-877-572-5511 | ENRICH@emory.edu | Emory University School of Medicine; Gustavo Pradilla, MD, Principal Investigator — 1-877-572-5511 | ENRICH@emory.edu | Emory University School of Medicine; Jonathan Ratcliff, MD, MPH, Principal Investigator — 1-877-572-5511 | ENRICH@emory.edu | Emory University School of Medicine
Locations (36):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute (BNI), Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Southern California (USC), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Delray Medical Center, Delray Beach, Florida
  - Baptist Health Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami / Jackson Memorial Hospital, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Vincent Indianapolis, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Saint Louis University, St Louis, Missouri
  - Washington University (Barnes Jewish), St Louis, Missouri
  - Cooper University Health Care, Camden, New Jersey
  - Albany Medical Center, Albany, New York
  - State University of New York, Buffalo, Buffalo, New York
  - New York Presbyterian Queens, Flushing, New York
  - Weill Cornell Medicine, New York, New York
  - Montefiore, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Geisinger Health System, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labib MA, Shah M, Kassam AB, Young R, Zucker L, Maioriello A, Britz G, Agbi C, Day JD, Gallia G, Kerr R, Pradilla G, Rovin R, Kulwin C, Bailes J. The Safety and Feasibility of Image-Guided BrainPath-Mediated Transsulcul Hematoma Evacuation: A Multicenter Study. Neurosurgery. 2017 Apr 1;80(4):515-524. doi: 10.1227/NEU.0000000000001316. PMID 27322807
- [Background] Chen CJ, Caruso J, Starke RM, Ding D, Buell T, Crowley RW, Liu KC. Endoport-Assisted Microsurgical Treatment of a Ruptured Periventricular Aneurysm. Case Rep Neurol Med. 2016;2016:8654262. doi: 10.1155/2016/8654262. Epub 2016 Apr 19. PMID 27195160
- [Background] Amenta PS, Dumont AS, Medel R. Resection of a left posterolateral thalamic cavernoma with the Nico BrainPath sheath: case report, technical note, and review of the literature. Interdisciplinary Neurosurgery: Advanced Techniques and Case Management. 2016; 5:12-17.
- [Background] Bauer AM, Rasmussen PA, Bain MD. Initial Single-Center Technical Experience With the BrainPath System for Acute Intracerebral Hemorrhage Evacuation. Oper Neurosurg. 2017 Feb 1;13(1):69-76. doi: 10.1227/NEU.0000000000001258. PMID 28931255
- [Background] Ziai W, Nyquist P, Hanley DF. Surgical Strategies for Spontaneous Intracerebral Hemorrhage. Semin Neurol. 2016 Jun;36(3):261-8. doi: 10.1055/s-0036-1582131. Epub 2016 May 23. PMID 27214701
- [Background] Fiorella D, Arthur A, Bain M, Mocco J. Minimally Invasive Surgery for Intracerebral and Intraventricular Hemorrhage: Rationale, Review of Existing Data and Emerging Technologies. Stroke. 2016 May;47(5):1399-406. doi: 10.1161/STROKEAHA.115.011415. Epub 2016 Apr 5. No abstract available. PMID 27048700
- [Background] Chen JW, Paff MR, Abrams-Alexandru D, Kaloostian SW. Decreasing the Cerebral Edema Associated with Traumatic Intracerebral Hemorrhages: Use of a Minimally Invasive Technique. Acta Neurochir Suppl. 2016;121:279-84. doi: 10.1007/978-3-319-18497-5_48. PMID 26463961
- [Background] Przybylowski CJ, Ding D, Starke RM, Webster Crowley R, Liu KC. Endoport-assisted surgery for the management of spontaneous intracerebral hemorrhage. J Clin Neurosci. 2015 Nov;22(11):1727-32. doi: 10.1016/j.jocn.2015.05.015. Epub 2015 Jul 31. PMID 26238692
- [Background] Ding D, Przybylowski CJ, Starke RM, Sterling Street R, Tyree AE, Webster Crowley R, Liu KC. A minimally invasive anterior skull base approach for evacuation of a basal ganglia hemorrhage. J Clin Neurosci. 2015 Nov;22(11):1816-9. doi: 10.1016/j.jocn.2015.03.052. Epub 2015 Jun 30. PMID 26142050
- [Background] Kassam AB, Labib MA, Bafaquh M, et al. Part II: an evaluation of an integrated systems approach using diffusion-weighted, image-guided, Exoscopic-assisted, transulcal radial corridors. Innovative Neurosurg. 2015; 3(1-2): 25-33.
- [Background] Kassam AB, Labib MA, Bafaquh M, et al. Part I: the challenge of functional preservation: an integrated systems approach using diffusion-weighted, image-guided, Exoscopic-assisted, transulcal radial corridors. Innovative Neurosurgy. 2015; 3(1-2): 5-23.
- [Background] Ritsma B, Kassam A, Dowlatshahi D, Nguyen T, Stotts G. Minimally Invasive Subcortical Parafascicular Transsulcal Access for Clot Evacuation (Mi SPACE) for Intracerebral Hemorrhage. Case Rep Neurol Med. 2014;2014:102307. doi: 10.1155/2014/102307. Epub 2014 Aug 6. PMID 25165588
- [Background] Zucker, L. Corticospinal tract restoration post parafascicular transulcal subcortical (thalamic) ICH evacuation. Poster #1450 presented at: 2016 Congress of Neurological Surgeons Annual Meeting; September 24-28, 2016; San Diego, CA.
- [Background] Chen J, Tran K, Dastur C, Stradling D, Yu W. The use of the BrainPath stereotactic guided surgery for the removal of spontaneous intracerebral hemorrhage: a single institutional experience. Abstract presented at: 2015 NeuroCritical Care Society Meeting; October 7-10, 2015; Scottsdale, AZ.
- [Background] Kulwin C, Rodgers R, Shah M. Preliminary experience with evacuation of intracerebral hemorrhage via a minimally invasive parafascicular technique. Presented at: 2015 Neurosurgical Society of America Annual Meeting; April 2015.
- [Background] Chen J, Kaloostian SW. Use of minimally invasive techniques under austere circumstances for the urgent resection of subcortical intracerebral hemorrhages. Poster #0075 presented at: 12th Annual Conference of the Society for Brain Mapping and Therapeutics; March 6-8, 2015.
- [Background] Britz G, Kassam AB, Labib M, Young R, Zucker L, Maioriello A, et al. Minimally invasive subcortical parafascicular access for clot evacuation: a paradigm shift. Poster # MP120 presented at: 2015 International Stroke Conference; February 11-13, 2015; Nashville, TN.
- [Background] Labib M, Britz G, Young R, Zucker L, Shah M, Kulwin CG, et al. The safety and efficacy of image-guided trans-sulcal radial corridors for hematoma evacuation: a multicenter study. Late breaking oral presentation LB12 at: 2015 International Stroke Conference; February 11-13, 2015; Nashville, TN.
- [Background] Kulwin CG, Shah MV. Minimally invasive parafascicular approach to deep cerebral lesions: initial Indiana University experience. Presented at: 2014 Neurosurgical Society of America Annual Meeting; June 2014.
- [Background] Labib M, Ghinda D, Bafaquh M, Kumar R, Agbi C, Kassam AB. The diffusion tensor imaging (DTI) guided Transulcul Exoscopic radial corridor approach for the resection of lesions in the sensorimotor area. Poster #1598 presented at: 2013 Congress of Neurological Surgeons Annual Meeting; October 19-23, 2013; San Francisco, CA.
- [Background] Ghinda DC, Bafaquh M, Labib M, Kumar R, Agbi CB, Kassam AB. A Transulcul Exoscopic radial corridor approach for the management of primary intracranial hemorrhage. Poster #1621 presented at: 2013 Congress of Neurological Surgeons Annual Meeting; October 19-23, 2013; San Francisco, CA.
- [Derived] Hanmer J, Arnold J, Hall A, Ratcliff JJ, Allen JW, Frankel M, Wright DW, Barrow DL, Pradilla G, Smith KJ; ENRICH Trial Investigators. Cost-Effectiveness Analysis of Early Minimally Invasive Removal of Intracerebral Hemorrhage. Stroke. 2025 Jul;56(7):1799-1806. doi: 10.1161/STROKEAHA.124.048493. Epub 2025 Apr 25. PMID 40276867
- [Derived] Pradilla G, Ratcliff JJ, Hall AJ, Saville BR, Allen JW, Paulon G, McGlothlin A, Lewis RJ, Fitzgerald M, Caveney AF, Li XT, Bain M, Gomes J, Jankowitz B, Zenonos G, Molyneaux BJ, Davies J, Siddiqui A, Chicoine MR, Keyrouz SG, Grossberg JA, Shah MV, Singh R, Bohnstedt BN, Frankel M, Wright DW, Barrow DL; ENRICH trial investigators; ENRICH Trial Investigators. Trial of Early Minimally Invasive Removal of Intracerebral Hemorrhage. N Engl J Med. 2024 Apr 11;390(14):1277-1289. doi: 10.1056/NEJMoa2308440. PMID 38598795
- [Derived] Ratcliff JJ, Hall AJ, Porto E, Saville BR, Lewis RJ, Allen JW, Frankel M, Wright DW, Barrow DL, Pradilla G. Early Minimally Invasive Removal of Intracerebral Hemorrhage (ENRICH): Study protocol for a multi-centered two-arm randomized adaptive trial. Front Neurol. 2023 Mar 16;14:1126958. doi: 10.3389/fneur.2023.1126958. eCollection 2023. PMID 37006503